CLINICAL TRIAL: NCT03160417
Title: Doppler Ultrasound in Rewarming After Targeted Control Management in Cardiac Arrest
Acronym: DTCHT
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: DTCHT
Record Dates: First submitted 2017-05-15; First posted 2017-05-19 (Actual); Last update posted 2022-09-07 (Actual); Status verified 2022-09

CONDITIONS: Cardiac Arrest; Doppler Ultrasound
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the study is to describe CBF modifications during rewarming after targeted temperature management in cardiac arrest patients

ELIGIBILITY:
Inclusion Criteria:

Major Cardiac arrest Targeted temperature management

Exclusion Criteria:

GCS>8 after cardiac arrest Neurologic cause of cardiac arrest

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cardiac arrest with GCS<8
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2016-04-25 (Actual); Primary Completion 2017-10-28 (Actual); Study Completion 2017-10-28 (Actual)

PRIMARY OUTCOMES:
Changes in TCD estimates of CBF measurements | day 3

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU Brest, Brest, Finistère, France